CLINICAL TRIAL: NCT04521335
Title: A Phase I Study of Disulfiram and Copper Gluconate in Patients With Treatment-Refractory Multiple Myeloma
Brief Title: Study of Disulfiram and Copper Gluconate in Patients With Treatment-Refractory Multiple Myeloma
Acronym: Repurpose-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed at PI's Request
Sponsor: University of Utah (Other)
Collaborators: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI131966
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Disulfiram; Gluconates

STUDY DESIGN:
Intervention Model Description: A standard 3+3 dose escalation design will be used to determine the recommended phase 2 dose (RP2D) while ensuring the safety and tolerability of the treatment. Once the RP2D has been assigned in dose-escalation, an expansion cohort will open to the enrollment of 14 additional patients to further characterize the safety and tolerability of the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): disulfiram and copper gluconate in combination
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate

INTERVENTIONS:
Drug: Disulfiram — Patients will be instructed to self-administer disulfiram and copper gluconate twice daily at the assigned dose level. Both medications will be administered in 28-day cycles.
Drug: Copper Gluconate — Patients will be instructed to self-administer disulfiram and copper gluconate twice daily at the assigned dose level. Both medications will be administered in 28-day cycles.

SUMMARY:
This is a phase I, open-label trial of disulfiram in combination with copper gluconate in patients with treatment-refractory multiple myeloma. The trial is designed to assess the Phase 2 Recommended Dose (RP2D) of disulfiram and copper gluconate in combination. The trial will open with dose escalation, followed to an expansion cohort to further characterize the safety and tolerance of the combination.

Dose escalation will utilize a standard 3+3 design and will test up to five dose levels. Dose levels will be separated into two sequential parts defined by the fixed dose of copper as copper gluconate administered with ascending doses of disulfiram. Part 1 of dose escalation will consist of dose levels 0 and 1 with the option to reduce to Dose Level -1 if Dose Level 0 is deemed intolerable. Part 2 will test dose levels 2 and 3. The Dose Level deemed to be the RP2D will be used in dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Relapsed or refractory myeloma that fits or did fit IMWG diagnostic criteria1 for symptomatic myeloma (although new or worsening end organ damage is not required to be eligible) as defined below:

  * Presence of > 10% clonal bone marrow plasma cells and/or biopsy-proven extramedullary plasmacytoma;
  * Evidence of myeloma defining event(s) attributed to the patient's myeloma:

    * Hypercalcemia: Serum calcium > 11.5 mg/dL; or
    * Renal Insufficiency: Serum creatinine > 2 mg/dL; or
    * Anemia > 2 g/dL below the lower limit of normal or hemoglobin value < 10 g/dL; or
    * Bone lesions: lytic lesions, severe osteopenia, pathologic fractures, or > 1 lesion on MRI at least 5 mm in size;
  * Bone marrow plasma cells > 60%
  * Serum free light chain ratio > 100
* Expansion cohort only: patients must have measurable disease defined as any of the following:

  * Serum monoclonal protein > 500 mg/dL by protein electrophoresis;
  * 200 mg of monoclonal protein in the urine on screening 24-hour electrophoresis;
  * Serum immunoglobulin free light chain > 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio.
* Progressed during or after an immunomodulatory drug, proteasome inhibitor, and anti-CD38 antibody, and at least 2 prior lines of therapy.
* ECOG performance status ≤ 2 or Karnofsky ≥ 60% (Appendix 1). --Note: Patients with lower performance status based solely on symptoms secondary to multiple myeloma are eligible.
* Adequate organ function as defined as:

  --Hematologic:
  * ANC ≥ 1000 /μL
  * Platelet count > 50,000 /μL

    --Hepatic:
  * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
* Normal serum copper levels and serum ceruloplasmin > 17 mg/dL.
* No known allergy to disulfiram or copper.
* Willing to refrain from ingestion of alcoholic beverages while in the study.
* Negative serum or urine pregnancy test at screening for women of childbearing potential ≤ 14 days prior to cycle one day one.
* Highly effective contraception for both male and female subjects throughout the study and for at least 14 days after last study treatment administration if the risk of conception exists.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior autologous and/or allogeneic transplant and/or CAR-T cell occurred ≤ 90 days prior to registration.
* Prior chemotherapy ≤ 2 weeks prior to the first dose of study treatment.
* Requires systemic corticosteroid therapy > 10 mg daily of prednisone or its equivalent for the management of symptoms or comorbid conditions.

  --Note: Doses of corticosteroid should be ≤ 10 mg prednisone or equivalent and stable for at least 7 days prior to starting study treatment to be deemed eligible.
* Receiving any other therapeutic investigational agents.
* Active treatment with any herbal or dietary supplements
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  --Cardiovascular disorders:
  * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before the first dose.
  * Left ventricular ejection fraction < 45% (only to be assessed at screening if clinically indicated).
* History of seizures, psychosis, or schizophrenia.
* History of liver disease, Wilson's disease, or hemochromatosis.
* Known HIV infection with a detectable viral load at the time of screening.

  --Note: Patients on effective antiretroviral therapy with an undetectable viral load at the time of screening are eligible for this trial.
* Active or ongoing infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes (POEMS) syndrome.
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug.
* Live attenuated vaccinations within ≤ 4 weeks of the first dose of study therapy.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3) including a history of rubber contact dermatitis for hypersensitivity to thiuram derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) during the DLT evaluation period. | time from cycle one day one until cycle two day one (28 days)
  assess the recommended phase 2 dose of disulfiram in combination with copper as copper gluconate in subjects with relapse/refractory multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sborov, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saifi MA, Shaikh AS, Kaki VR, Godugu C. Disulfiram prevents collagen crosslinking and inhibits renal fibrosis by inhibiting lysyl oxidase enzymes. J Cell Physiol. 2022 May;237(5):2516-2527. doi: 10.1002/jcp.30717. Epub 2022 Mar 13. PMID 35285015